CLINICAL TRIAL: NCT04982432
Title: Orismilast for the Treatment of Mild to Severe Hidradenitis Suppurativa (OSIRIS)
Brief Title: Orismilast for the Treatment of Mild to Severe Hidradenitis Suppurativa
Acronym: OSIRIS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gregor Jemec (Other)
Collaborators: UNION therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Gregor Jemec, Professor, Zealand University Hospital
Organization: Zealand University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSIRIS [UNI50007-201]; 2021-000049-42 (EudraCT Number)
Record Dates: First submitted 2021-07-26; First posted 2021-07-29 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Intervention Model Description: Patients will be graded and assigned to a severity group (mild, moderate, or severe). All groups will receive the same intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orismilast (Experimental): Orismilast tablet, oral administration, multiple titrated doses twice daily, 10 mg up to 40 mg, morning and evening, 16 weeks treatment.
  Interventions: Drug: Orismilast

INTERVENTIONS:
Drug: Orismilast — Orismilast is a next generation PD4 inhibitor with demonstrated broad anti inflammatory properties
  Other Names: UNI5001

SUMMARY:
The purpose of this study is to assess the efficacy and safety of oral administration of orismilast for treatment of mild, moderate, or severe hidradenitis suppurativa (HS) in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult patients, 18 years of age or older.
2. Have mild to severe HS for at least 1 year prior to the baseline visit, as determined by the investigator through participant interview and/or review of the medical history.
3. Have HS lesions in at least 2 distinct anatomic area (right/left axillary, inguinal, inframammary, abdominal, perineal).
4. Has a total inflammatory lesions (AN) count of greater than or equal to 2.
5. Total draining fistula count of less than or equal to 30.
6. A stable analgesic dose for 2 weeks prior to baseline.

Exclusion Criteria:

1. Presence of active skin lesions other than HS that could interfere with the assessment of HS.
2. Receipt of prescription topical therapies for HS within 7 days prior to the baseline visit (Visit 2).
3. Receipt of systemic therapies for HS, within 28 days prior to the baseline visit.
4. Any oral antibiotic within 28 days prior to baseline visit.
5. Receipt of a live vaccine within 14 days prior to screening.
6. Biologic use for indications other than HS within a minimum of 30 days or 5 half-lives of the drug, whichever is longer, prior to baseline.
7. Treatment with any investigational drug of chemical or biologic nature within a minimum of 30 days or 5 half-lives of the drug, whichever is longer, prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent change from Baseline in AN (abscesses and nodules) count at Week 16 | Day 1 to Week 16
  Total count of abscess and inflammatory nodules

SECONDARY OUTCOMES:
Change from Baseline in abscess, nodule, and draining fistula counts at Week 16 | Day 1 to Week 16
  Total count of abscess, inflammatory nodules, and draining fistula
Change from Baseline in IHS4 value at Week 16 | Day 1 to Week 16
  ISH4 is a validated international clinimetric scale. The score is based on a count of inflamed lesions. The resulting IHS4 score is arrived at by the number of nodules (multiplied by 1) plus the number of abscesses (multiplied by 2) plus the number of draining tunnels (multiplied by 4).
Change from Baseline in Patient's Global Assessment of Skin Pain (NRS) at Week 16 | Day 1 to Week 16
  Completion of questionnaire covering skin pain Patient's Global Assessment of Skin Pain (0=no pain, 10=worst imaginable pain) 0-10 Numerical Rating Scale (NRS).
Change from Baseline in HiSQOL Total Score at Week 16 | Change from Baseline in HiSQOL Total Score at Week 16
  Patient completion of the Hidradenitis Suppurativa Quality of Life (HiSQOL) questionnaire that contains Hidradenitis Suppurativa specific items such as drainage and odor in addition to more general skin specific items

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Jemec, Professor, Principal Investigator — Zealand University Hospital

IPD SHARING:
Plan to Share IPD: No